CLINICAL TRIAL: NCT07240935
Title: Validation of the Spanish Version of a Psychosocial Needs Assessment Questionnaire for Adolescents and Young Adults With Cancer (AYA-POST)
Brief Title: Spanish Validation of a Psychosocial Needs Assessment for Adolescents and Young Adults With Cancer (AYA-POST)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PR(AMI)132/2025
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: AYA Cancer Patients
Keywords: AYA cancer psychosocial; AYA cancer Distress Thermometer; AYA cancer psychosocial needs

STUDY DESIGN:
Intervention Model Description: Interventional: Participants only will complete the psychosocial scales and QoL, but none other intervention would be done and treatmentand supportive care will remain the same for participants and non participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYA-POST Spanish (Experimental)
  Interventions: Other: AYA-POST questionaries

INTERVENTIONS:
Other: AYA-POST questionaries — AYA-POST questionaries includes: Distress Thermometer and psychosocial needs assesment

SUMMARY:
This prospective multicenter study aims to validate the Spanish version of the Distress Thermometer and accompanying list of psychosocial needs specifically adapted for adolescents and young adults (AYA) aged 15 to 25 who are diagnosed with cancer.

These tools, firstly developed by the National Comprehensive Cancer Network (NCCN) and then specifically adapted for AYA by Canteen Australia and validated in English-speaking countries, are widely used around the world to quickly identify emotional distress and unmet practical or social needs in cancer patients, helpting to detect their emotional distress and support needs, which can differ significantly from those of children or older adults.

By validating these screening tools in Spanish this study seeks to confirm whether they can reliably identify young patients who may be experiencing psychosocial difficulties.

Once validated, these tools can be easily integrated into clinical practice in Spanish-speaking countries, helping healthcare teams quickly identify vulnerable young patients, respond to their emotional needs earlier, and improve the overall quality of care.

The results will also highlight which psychosocial needs are most common in AYA cancer patients, supporting the development of future programs and services tailored to this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 15 and 25 years old who provide informed consent (> 18 yo) or parents informed consent and patient consent in case of minors (15 to 18 yo)
* Diagnosis of cancer (malignant solid tumor or hematologic malignancy) within 6 months prior to study inclusion or whose first non-surgical treatment (chemotherapy, radiotherapy, or targeted therapy) started within the last 6 months.
* Treated from diagnosis or first non-surgical treatment at centers where the study is open.

Exclusion Criteria:

* Patients who are not receiving their first line of non-surgical treatment.
* Patients who do not have good understanding of Spanish (language used for the screening tool and questionnaires).
* Patients with severe neurological impairment or other conditions that, in the investigator's opinion, prevent proper completion of study procedures.

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2031-10-31 (Estimated); Study Completion 2032-10-31 (Estimated)

PRIMARY OUTCOMES:
Validation of the Spanish version of AYA-POST | From enrollment to the end of follow-up 1 year after finishing cancer treatment
  Correlation between the Spanish AYA-POST and currently validated HADS

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall Hebron, Barcelona, Barcelona, Spain